CLINICAL TRIAL: NCT06283914
Title: Imputation of Arterial Oxygen Partial Pressures Using Pulse Oximetry in Surgical Patients Under General Anesthesia
Brief Title: Imputation of Arterial Oxygen Partial Pressures Using Pulse Oximetry
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Marwan Rizk, Principal Investigator, American University of Beirut Medical Center
Other Study IDs: BIO-2024-0011
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Oxygen Saturation; Respiratory Distress Syndrome; Anesthesia, General
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to validate existing PaO₂ prediction equations (Rice, Pandharipande, Gadrey, Hill, Severinghaus-Ellis) by comparing predicted PaO₂ values with measured values. If these equations are found to be invalid, new PaO₂ prediction formulas will be derived and validated for accuracy and performance.

The included blood samples are arterial blood sample collected for ABGs analysis through either an arterial catheter or an arterial blood puncture in adult patients (Age >18 years) undergoing general anesthesia regardless of the acuity of the surgery (elective, emergency, or lifesaving), the hemodynamic stability of the patient, or the comorbidities. Patients undergoing cardiac or thoracic surgeries will be excluded.

DETAILED DESCRIPTION:
The partial pressure of oxygen in the arterial blood (PaO2) / the fraction of inspired oxygen (FiO2) ratio has been commonly used as an indicator of adequate oxygenation and in the diagnosis and severity of acute respiratory distress syndrome (ARDS) which requires arterial blood gas (ABGs) analysis. Another way to measure oxygenation is by using the noninvasive pulse oximetry to measure the oxygen saturation (SpO2). Three formulas have been derived and validated in the intensive care unit (ICU) setting to estimate the PaO2 from the SpO2. However, the relationship of PaO2 and SpO2 and these derivation equations are not validated in the setting of general anesthesia in the operating theatre (OT) in which patients are prone to multiple intraoperative and postoperative pulmonary complications.

The aim is to validate existing PaO₂ prediction equations (Rice, Pandharipande, Gadrey, Hill, Severinghaus-Ellis) by comparing predicted PaO₂ values with measured values. If these equations are found to be invalid, new PaO₂ prediction formulas will be derived and validated for accuracy and performance.

This is a prospective cohort study that will be conducted at the American University of Beirut Medical Center (AUBMC) in the OT under the Department of Anesthesiology and Pain Medicine. The data will be collected by the investigators of the study. These include the PaO2 (in mmHg), FiO2, SpO2 (in %), and Mean airway pressure (in cmH2O) at the time of sample collection, in addition to patient characteristics as age, gender, weight, height, BMI, smoking status, surgery type, surgery acuity, and present comorbidities specifically cardiac and respiratory comorbidities.

Validating the use of one of the formulas to derive PaO2 from SpO2 in the OT would help anesthesiologists detect derangements in patients' oxygenation earlier and decrease the need for ABGs analysis and its possible complications.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Undergoing general anesthesia

Exclusion Criteria:

* Patients undergoing cardiac or thoracic surgeries will be excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The included blood samples are arterial blood sample collected for ABGs analysis through either an arterial catheter or an arterial blood puncture in adult patients (Age >18 years) undergoing general anesthesia regardless of the acuity of the surgery (elective, emergency, or lifesaving), the hemodynamic stability of the patient, or the comorbidities. Patients undergoing cardiac or thoracic surgeries will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
PaO2 | 30 minutes after intubation until extubation
  Partial pressure of oxygen in the arterial blood (PaO2)

OTHER OUTCOMES:
SpO2 | 30 minutes after intubation until extubation
  oxygen saturation (SpO2)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Rizk, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No